CLINICAL TRIAL: NCT04216199
Title: Role of Point of Care Ultrasound in Confirmation of Endotracheal Tube Placement in Children
Brief Title: Role of Point of Care Ultrasound in Endotracheal Tube Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: elbahnasawy
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Endotracheal Tube Wrongly Placed During Anesthetic Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Point of care Ultrasound (Experimental): Point of care Ultrasound for placement of endotracheal tube
  Interventions: Device: Point of care Ultrasound
- Traditional (No Intervention): Traditional method of insertion of endotracheal tube

INTERVENTIONS:
Device: Point of care Ultrasound — Point of care Ultrasound
  Other Names: POC Ultrasound
  Arms: Point of care Ultrasound

SUMMARY:
Role of point of care ultrasound in endotracheal tube placement in children

DETAILED DESCRIPTION:
Role of point of care ultrasound in confirmation of endotracheal tube placement in children

ELIGIBILITY:
Inclusion Criteria:

* Children below 18 years needing endotracheal intubation.

Exclusion Criteria:

* Age more than 18 years.
* Patients with significant neck or lung pathology.
* Patients with elective intubation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-20 (Estimated)

PRIMARY OUTCOMES:
Number of patients with correct placement of endotracheal tube | 6 months
  The number of patients with correct placement of endotracheal tube

CONTACTS AND LOCATIONS:
Overall Officials: Fekry khater, Msc, Principal Investigator — Emergency medicine department - Alazhar University; Mohamed S Sharaf, Prof., Principal Investigator — Anasthesia and Pain department - Alazhar University; Mohamed H Elshafey, Prof, Study Director — Radiodiagnosis Department - Tanta University; Mohamed G Elbahnasawy, Lecturer, Study Director — Emergency medicine department - Tanta University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No